CLINICAL TRIAL: NCT05904171
Title: Cognitive, Affective, and Motor Effects of Tangotherapy in Parkinson's Disease
Acronym: TANGOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25C304
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Argentine Tango; Dance Therapy; Cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangotherapy (Experimental): 2 hours of group-based Tangotherapy, weekly, for 6 weeks
  Interventions: Behavioral: Tangotherapy
- Physical Activity (Active Comparator): 2 hours of group-based physical activity, weekly, for 6 weeks
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Tangotherapy — Learning and practicing a series of moves - both individual and with a partner - taken from Argentine Tango, according to the Riabilitango (R) approach. The training is aimed at improving both physical (e.g., balance, change of direction, coordination, endurance) and cognitive (i.e., learning, divided attention, inhibition, planning) domains, in a pleasant, enjoyable, and inclusive environment.
  This group-based training will take place twice a week (1h each session), for 6 weeks.
  Arms: Tangotherapy
Behavioral: Physical activity — Walking and stretching in group twice a week (1h each session), for 6 weeks.
  Arms: Physical Activity

SUMMARY:
Neuroscientific research has shown a close relationship between physical fitness and cognition, showing a positive effect of physical activity (e.g., aerobic activity) on the maintenance of psycho-cognitive well-being in the elderly. In particular, dancing seems to be very effective, as it involves both motor and multisensory aspects (touch, sight, hearing, proprioception), stimulating memory, motor learning and social interaction. In fact, dance increases sensory-motor skills and cognitive performance in the neurologically healthy elderly. Dance-based therapeutic approaches, in particular Argentine tango, have also been implemented in the context of neurodegenerative pathologies, including Parkinson's disease (PD) where motor (i.e., tremors, postural instability, motor slowdown) and cognitive difficulties (e.g., executive deficits) may coexist. Most of these studies have so far demonstrated a significant improvement in balance and a reduction in motor symptoms, while evidence regarding cognitive and emotional benefits brought about by dance remains limited. When investigated, cognitive benefits have often been evaluated at the level of global cognition (i.e., screening tests), without a detailed characterization of the effects of tango on cognitive and affective functioning (e.g., executive functions, social cognition, depressive symptoms), central aspects in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild-moderate Parkinson's Disease (modified Hoehn&Yahr Scale 1-3)

Exclusion Criteria:

* Having attended Argentine Tango classes in the past year;
* Having attended Physical Therapy rehabilitation in the past month;
* Other neurological diseases (e.g., stroke, traumatic brain injury, brain tumors)
* Dementia
* Any clinical condition not compatible with physical activity
* Deep Brain Stimulation of infusion pumps implants

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Parkinson's Disease Cognitive Rating Scale (PD-CRS) - total score | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A battery of cognitive tests of memory, selective attention, visuo-spatial skills, and flexibility.
Change in Hospital Anxiety and Depression Scale (HADS) - total score | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A scale assessing depressive and anxiety symptoms.
Change in Health-related quality of Life (EQ-5D-5L) - total score | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A questionnaire about quality of life in different health-related domains.
Change in Stroop Task - reading time | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A test assessing cognitive inhibition.
Change in 6 minutes walking Test (6MWT) - Distance Walked | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A test assessing walking performance; i.e., distance walked in 6 minutes.
Change in Timed Up and Go (TUG) test - Execution Time | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A test used to assess a person's mobility.
Change in 10 meters walking test (10mWT) - Execution Time | At the beginning of the treatment, at the end of the treatment (i.e., after 6 weeks), and at 45 days follow-up
  A test assessing walking performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Bolognini, PhD, Principal Investigator — Laboratorio di Neuropsicologia, IRCCS Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
individual data will be uploaded on zenodo.com

REFERENCES:
- [Background] Carvalho A, Rea IM, Parimon T, Cusack BJ. Physical activity and cognitive function in individuals over 60 years of age: a systematic review. Clin Interv Aging. 2014 Apr 12;9:661-82. doi: 10.2147/CIA.S55520. eCollection 2014. PMID 24748784
- [Background] Kattenstroth JC, Kalisch T, Holt S, Tegenthoff M, Dinse HR. Six months of dance intervention enhances postural, sensorimotor, and cognitive performance in elderly without affecting cardio-respiratory functions. Front Aging Neurosci. 2013 Feb 26;5:5. doi: 10.3389/fnagi.2013.00005. eCollection 2013. PMID 23447455
- [Background] Kattenstroth JC, Kolankowska I, Kalisch T, Dinse HR. Superior sensory, motor, and cognitive performance in elderly individuals with multi-year dancing activities. Front Aging Neurosci. 2010 Jul 21;2:31. doi: 10.3389/fnagi.2010.00031. eCollection 2010. PMID 20725636
- [Background] Ismail SR, Lee SWH, Merom D, Megat Kamaruddin PSN, Chong MS, Ong T, Lai NM. Evidence of disease severity, cognitive and physical outcomes of dance interventions for persons with Parkinson's Disease: a systematic review and meta-analysis. BMC Geriatr. 2021 Sep 22;21(1):503. doi: 10.1186/s12877-021-02446-w. PMID 34551722
- [Background] Duncan RP, Earhart GM. Randomized controlled trial of community-based dancing to modify disease progression in Parkinson disease. Neurorehabil Neural Repair. 2012 Feb;26(2):132-43. doi: 10.1177/1545968311421614. Epub 2011 Sep 29. PMID 21959675
- [Background] Rios Romenets S, Anang J, Fereshtehnejad SM, Pelletier A, Postuma R. Tango for treatment of motor and non-motor manifestations in Parkinson's disease: a randomized control study. Complement Ther Med. 2015 Apr;23(2):175-84. doi: 10.1016/j.ctim.2015.01.015. Epub 2015 Feb 9. PMID 25847555
- [Derived] Caronni A, Amadei M, Diana L, Sangalli G, Scarano S, Perucca L, Rota V, Bolognini N. In Parkinson's disease, dual-tasking reduces gait smoothness during the straight-walking and turning-while-walking phases of the Timed Up and Go test. BMC Sports Sci Med Rehabil. 2025 Mar 7;17(1):42. doi: 10.1186/s13102-025-01068-8. PMID 40055732